CLINICAL TRIAL: NCT03651401
Title: Scapular Muscle Endurance, Shoulder Pain, and Functionality in Patients With Rotator Cuff Related Shoulder Pain: A Matched, Case-Control Study
Brief Title: Scapular Muscle Endurance, Shoulder Pain, and Functionality
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ugur Sozlu, Research assistant, Gazi University
Other Study IDs: 25901600-577
Record Dates: First submitted 2018-08-26; First posted 2018-08-29 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Rotator Cuff Syndrome of Shoulder and Allied Disorders
Keywords: Scapula; Endurance; Disability; Rotator cuff lesions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rotator cuff related shoulder pain: Participants were assessed for SME, pain (rest, activity, night, measurement), and upper extremity function (FIT-HaNSA).
  Interventions: Device: Scapular muscle endurance test; Other: Pain intensity; Device: Upper Limb Functional Performance
- age gender matched healthy controls: Participants were assessed for SME, and upper extremity function (FIT-HaNSA).
  Interventions: Device: Scapular muscle endurance test; Device: Upper Limb Functional Performance

INTERVENTIONS:
Device: Scapular muscle endurance test — The SME test, developed by Edmondston et al. 17, is based on an exercise used to improve the performance of the serratus anterior and trapezius muscles. The test was carried out while the subjects were facing the wall in standing position and with their shoulders and elbows flexed to 90 degrees. While both scapulae were in neutral position, an appropriate size of stick (18-36 cm) was selected and placed between the elbows, and they were asked to hold the dynamometer (Feta 137 F0202 1 kg/10 N) between their hands.
Other: Pain intensity — Pain intensity assessment was performed by questioning rest, activity, night, and measuremant pain using a visual analogue scale (VAS) on a 10 cm line with marks at both ends to define the limits of the pain experience as "no pain" (0) and "maximum pain experienced" (10), with higher scores indicating greater pain 20.
  Groups: rotator cuff related shoulder pain
Device: Upper Limb Functional Performance — The Functional Impairment Test-Hand and Neck/Shoulder/Arm (FIT-HaNSA) protocol, which was developed by MacDermid et al. 21, was used to evaluate the functional performance of the upper extremity when performing 3 tasks.
  Other Names: FIT-HaNSA

SUMMARY:
The purpose of this study is to compare scapular muscle endurance (SME), shoulder pain, and functionality of patients with rotator cuff related shoulder pain (RCRSP) with those in the age-gender matched healthy controls and to evaluate the relationship between SME with shoulder pain, and functional impairments in patients with RCRSP.

DETAILED DESCRIPTION:
Patients with RCRSP (n:23), and age-gender matched healthy controls (n:23) were included in the study. SME were measured by a one-kilogram dynamometer while the shoulder and elbows are flexed 90°. Self-reported pain intensity (activity, night, after SME and FIT-HaNSA) was assessed visual analog scale (VAS). Functionality was also assessed using the Functional Impairment test-hand, neck, shoulder, and arm (FIT-HaNSA).

ELIGIBILITY:
Inclusion criteria:

* Positive sign in two or more specific shoulder clinical tests;
* The presence of RCRSP in magnetic resonance imaging (MRI);
* At least 120° flexion, 25° abduction, and 30° external rotation movements of the shoulder;
* Being right arm dominant;
* No surgical history in the shoulder region.

Exclusion criteria:

* Patients with shoulder pathology other than RCRSP such as glenohumeral instability (capsular and ligamentous lesions, labral lesions, or bone lesions), bicipital tendon lesions, acromioclavicular joint osteoarthritis, glenohumeral joint osteoarthritis, adhesive capsulitis, shoulder or cervical surgery history,
* Neurological and systemic inflammatory diseases,
* Bilateral shoulder complaints,
* Cardiovascular system diseases,
* Pregnancy,
* Underwent shoulder-related physical therapy within the past three months.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 23 patients and 23 age-gender matched healthy subjects who met the inclusion criteria were included to the study
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Scapular muscle endurance | Baseline assessment, no follow-up
  Unit of Measure:second
Pain intensity | Baseline assessment, no follow-up
  Unit of Measure:visual analogue scale
Upper Limp Functional Performance | Baseline assessment, no follow-up
  Protocol: FIT-HaNSA

CONTACTS AND LOCATIONS:
Overall Officials: Selda BAŞAR, Study Chair — Gazi University

IPD SHARING:
Plan to Share IPD: No